CLINICAL TRIAL: NCT01668732
Title: Decision Making Deficit and DNA Methylation in Opioid Receptor Genes Among Community Heroin Addicts
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: MD101SCW01
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Heroin Addiction
MeSH Terms: conditions — Heroin Dependence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- community heroin addicts

SUMMARY:
Heroin addiction has emerged as a serious problem with tremendous impacts on the addicts and the society. Since the introduction of opioids substitutive treatment in 2006, more than 30,000 heroin addicts had received treatment, and nearly 12,000 continued on treatment currently. However, an unknown proportion of patients hidden in community remained un-treatment. To motivate the community heroin addicts is thus a challenging task.

It is suggested that decision making deficit is core feature which determine outcomes and treatment motivations in patients with addiction disorders. Recently, the state-of-the-art development of epigenetics uncover that environmental modification, via altering level of DNA methylation and gene expression will influence on neurocognitive functioning.

Via respondent-driven sampling, this study aims to recruit a representative sample targeting at the hard-to-reach community heroin addicts. The goal of this study is to identify the clinical feature as well as decision making-related neurocognitive deficit in these patients. Moreover, the investigators will explore the interplay of clinical features, DNA methylation and gene expressions on opioids receptor genes. The findings will help to clarify the clinical characteristics of community heroin addicts, to uncover the links between DNA methylation and clinical features of heroin addiction and to develop modifiable treatment targets in the future.

ELIGIBILITY:
Inclusion Criteria:

* 1) 20 to 65 of age; 2) meeting DSM-IV criteria of opioids dependence

Exclusion Criteria:

-

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community heroin addicts
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Chang Wang, M.D., M.Sc., Principal Investigator — National Health Research Institute, Taiwan